CLINICAL TRIAL: NCT01394367
Title: Study of Influence of Respiratory and Exercise Therapy on Oxygen Uptake, Quality of Life and Right Ventricular Function in Severe Pulmonary Hypertension
Brief Title: Influence of Respiratory and Exercise Therapy on Oxygen Uptake, Quality of Life and Right Ventricular Function in Severe Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S-472/2009
Record Dates: First submitted 2011-06-28; First posted 2011-07-14 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Hypertension
Keywords: respiratory therapy; exercise therapy; oxygen uptake; quality of life; right ventricular function; severe pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Respiratory Rate; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory and exercise therapy (Experimental): Randomized, prospective, controlled, blinded study of three-week inpatient rehabilitation and subsequent continuing of the training at home for 12 weeks. The control group received conventional rehabilitation without a specific training program. After 15 weeks training is also offered to patients in the control group.
  Interventions: Other: respiratory and exercise therapy
- respiratory and exercise therapy (No Intervention)

INTERVENTIONS:
Other: respiratory and exercise therapy — Conventional therapy with diet, massage, relaxation baths, plus easy strolls specific respiratory and physical therapy plus mental walking training

SUMMARY:
Aim of this study is to investigate whether and to what extent a cautious respiratory and exercise therapy can complement medical treatment and change the condition, oxygen uptake, quality of life, the pulmonary vascular pressures, the size of the right heart and the 6-minute walk distance in patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Consent form
* men and women> 18 years <75 years
* invasively confirmed chronic PH who have received complete diagnostic evaluation by specialized doctors / physicians according to the WHO classification at a center for pulmonary hypertension and were adjusted for 2 months under intensive medical therapy and are stable.

Exclusion Criteria:

* Pregnancy or lactation
* Change in medication during the last 2 months
* Patients with signs of right heart decompensation
* severe walking disturbance
* uncertain diagnoses
* No previous invasively confirmation of PH
* acute diseases, infections, fever
* Serious lung disease with FEV1 <50% or TLC <70% of target
* Further exclusion criteria are the following diseases: active myocarditis, unstable angina pectoris, exercise-induced ventricular arrhythmias, congestive heart failure, significant heart disease, pacemakers, and hypertrophic obstructive cardiomyopathy, or a highly reduced left ventricular function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Improvement of peak O2 uptake (VO2peak) under stress | up to 15 weeks
  Three-week inpatient rehabilitation, continuation of the training program for another 12 weeks at home (exercise group), patients in the control group continued their usual activities. After 15 weeks, training is also offered to patients in the control group.

SECONDARY OUTCOMES:
Changes in hemodynamics at rest and during exercise | up to 15 weeks
  1. Changes in hemodynamics at rest and during exercise after three weeks and 15 weeks: RAP, RVP, sPAP, DPAP, mPAP, PCWP, cardiac output, PVR, CI, SvO2
  2. Changes in exercise capacity: 6-minute walk distance, Recumbent Bike (Watts), respiratory economy (EQO2, EQCO2)
  3. Improved condition(NYHA class, Borg scale)
  4. Changes in MRI and echocardiographic parameters of right and left ventricle: size and pump function.
  5. Change of laboratory parameters, which are markers of right heart failure as NTproBNP, interleukins

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, Professor, Study Director — Center for pulmonary hypertension, Thoraxclinic Heidelberg
Locations (1):
- Center for pulmonary Hypertension, Thoraxclinic Heidelberg, Heidelberg, Germany